CLINICAL TRIAL: NCT05512962
Title: A Multi-Center, Randomized, Two-Arm, Parallel-Group, Single-masked, 24-week, Clinical Trial to Evaluate Safety and Tolerability of Two Dose Levels of Suprachoroidal Triamcinolone Acetonide Administered With the Oxulumis® Ophthalmic Administration Device in Subjects With Diabetic Macular Edema
Brief Title: Oxulumis® Suprachoroidal Microcatherization of Triesence® in Diabetic Macular Edema
Acronym: CAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxular Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OXUCT-103 - CAPE; 2022-001533-37 (EudraCT Number)
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Parallel Two-Dose Group Assignment
Who Masked: Participant
Masking Description: Subjects will be masked to the dose level of triamcinolone acetonide administered with the suprachoroidal Oxulumis® microcatheter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Suprachoroidal Triamcinolone acetonide 2.4mg (Experimental): The Oxulumis® device will be used for the administration of Triesence® (Triamcinolone acetonide) via suprachoroidal microcatheterization. A single treatment with 2.4mg/60µl Triesence® will be applied.
  Interventions: Drug: Triamcinolone Acetonide; Device: Semi-automated Suprachoroidal Microcatheter
- Suprachoroidal Triamcinolone acetonide 4.0mg (Experimental): The Oxulumis® device will be used for the administration of Triesence® (Triamcinolone acetonide) via suprachoroidal microcatheterization. A single treatment with 4.0mg/100µl Triesence® will be applied.
  Interventions: Drug: Triamcinolone Acetonide; Device: Semi-automated Suprachoroidal Microcatheter

INTERVENTIONS:
Drug: Triamcinolone Acetonide — Single suprachoroidal Administration of Triamcinolone acetonide
  Other Names: Triesence®
Device: Semi-automated Suprachoroidal Microcatheter — Ophthalmic Adminstration Device
  Other Names: Oxulumis®

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and tolerability of suprachoroidal microcatheterization with the Oxulumis® device for a randomized treatment with two dose levels of Triesence® in subjects with Diabetic Macular Edema.

DETAILED DESCRIPTION:
Twenty-four (24) week, randomized, two-arm, single-masked, clinical trial to evaluate safety, tolerability, and to explore the efficacy of two dose levels of suprachoroidal triamcinolone acetonide suspension (Triesence®, 2.4 mg, and 4.0mg) administered using the Oxulumis® microcatheterization device in subjects with previously treated Diabetic Macular Edema.

After a screening period, approximately 20 eligible Diabetic Macular Edema subjects will be treated using a 1:1 ratio to receive a single administration of one of two dose levels of triamcinolone acetonide (low dose, 2.4mg. or mid-dose, 4.0mg, respectively). If for any reasons treatment in randomized subjects cannot be completed, additional consecutive subjects will be randomized until the target number of approximately 20 treated subjects is reached.

From Week 4, subjects will be assessed for the need for follow-on treatment. The follow-up period after treatment administration will be up to twenty-four (24) weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes mellitus.
* Diabetic macular edema involving the center of the fovea in the study eye
* Best-corrected visual acuity in the study eye of ≤73 (early treatment of diabetic retinopathy study) ETDRS letters (approximate Snellen equivalent of 20/40 or worse)
* Short-lived, limited, or no response to prior ocular injection therapy

Exclusion Criteria:

* Macular edema is considered due to a cause other than diabetes mellitus in the study eye.
* Condition, in the study eye, in which visual acuity is not expected to improve from the resolution of macular edema
* Macular laser photocoagulation or panretinal laser photocoagulation in the study eye performed within sixteen (16) weeks prior to screening.
* Active proliferative diabetic retinopathy (PDR) or sequelae of PDR in the study eye.
* Active malignancy or history of malignancy within the past five years.
* Prior intravitreal (IVT) treatment with anti-Vascular endothelial growth factor (VEGF) in the study eye: last injection within four weeks, before screening
* Prior ocular treatment with steroids in the study eye: last injection (intra- or periocular) with triamcinolone acetonide within three (3) months, with dexamethasone implant (Ozurdex®) within six (6) months before screening.
* Prior treatment with longer duration steroid implants (e.g., fluocinolone acetonide IVT implant, Iluvien®) is exclusionary.
* Prior treatment with suprachoroidal steroids is exclusionary.
* Uncontrolled diabetes with a hemoglobin A1c (HbA1c) > 12% or any other uncontrolled systemic disease at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Asmus, MD, Study Director — Oxular Limited
Locations (6):
- United States (6):
  - California Retina Consultants, Bakersfield, California
  - Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas - The Woodlands, Houston, Texas
  - Retina Consultants of Texas - Bellaire, Houston, Texas
  - Retina Consultants of Texas - San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive recruitment at participating sites in the US. Enrolment will be continued, until at least 20 randomized subjects could also be treated, i.e. total enrolment could be higher than 20.
Period: Overall Study
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Started (= Safety Population of all eligible subjects randomized) | 13 | 12
Efficacy Evaluable Population (All subjects with completed administration of study treatment and at least 1 post baseline assessment) | 10 | 10
Per Protocol Population (EEP subjects without major protocol deviations impacting efficacy outcomes) | 5 | 9
Completed (Based on Efficacy Evaluable Population) | 12 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population (all subjects eligible and randomized)
Groups:
- Total: Total of all reporting groups
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (8.32) | 63.2 (6.78) | 63.0 (7.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
Diabetes Type [Count of Participants; unit: Participants]
  Type 1 | 1 | 0 | 1
  Type 2 | 12 | 12 | 24
Duration of Diabetes (years) [Mean (Full Range); unit: years] | 19.4 [1.3 to 45.1] | 20.3 [6.0 to 34.5] | 19.9 [1.3 to 45.1]
Duration of DME (years), mean (min-max) [Mean (Full Range); unit: years] | 2.7 [0.2 to 7.2] | 4.2 [0.5 to 9.1] | 3.4 [0.2 to 9.1]
Lens status, n (%) (Study Eye) [Number; unit: participants] — Clinical Examination, e.g. using a Slit Lamp to inspect the ocular lens. Categories are aphakic (no lens present), phakic (lens present), pseudophakic (artificial lens, typically after cataract surgery for lens replacement).
  participants
    Aphakic (no lens present) | 0 | 0 | 0
    Phakic (lens present) | 8 | 5 | 13
    Pseudophakic (artificial lens present) | 5 | 7 | 12
Central Subfield Thickness (Study Eye) [Mean (Standard Deviation); unit: µm] — assessed at the Baseline Visit before treatment Population: for the efficacy evaluable population with completed administration of trial treatment
  µm | 530.2 (128.2) | 560.4 (166.8) | 544.7 (145.7)
ETDRS BCVA, mean (SD) (Study Eye) [Mean (Standard Deviation); unit: ETDRS letters] — based on duplicate assessment of BCVA at the respective visit, here the Baseline Visit before treatment Population: for the Efficacy Evaluable Population with completed administration of trial treatment
  ETDRS letters | 60.9 (12.4) | 52.9 (14.2) | 57.1 (13.7)
IOP (mmHg), mean (SD) (Study Eye) [Mean (Standard Deviation); unit: mmHg] — assessed at the Baseline Visit before treatment
  mmHg | 16.2 (3.11) | 16.1 (3.34) | 16.1 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Ocular Adverse Events, Systemic Adverse Events, Serious, and Treatment-emergent Non-serious Adverse Events
Description: Treatment-emergent ocular adverse events are defined as an ocular event that emerges following the start of administration of Triesence® with the Oxulumis® microcatheter at Visit 2 (Baseline, Day 0)
Time Frame: Day 0 up to Week 24 (per protocol individual trial duration per participant)
Population: Safety Analysis set of subjects enrolled - Number of Patients with at least 1 event
Measure: Count of Participants; unit: Participants
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 13 | 12
Participants
  Number of Participants with Ocular Treatment-Emergent Adverse Events | 10 | 8
  Number of Participants with Systemic (Non-Ocular) Treatment-Emergent Adverse Events | 3 | 5
  Number of Participants with Ocular Treatment-Emergent Serious Adverse Events | 0 | 0
  Number of Participants with Systemic (Non-Ocular) Treatment-Emergent Serious Adverse Events | 0 | 0

2. Primary Outcome: Frequency of Adverse Device Effects and Frequency of Serious Adverse Device Effects
Description: Adverse device effects a are defined as effects that emerge following the start of administration of the Oxulumis® microcatheter at Visit 2 (Baseline, Day 0)
Time Frame: Day 0 up to Week 24 (per protocol individual trial duration per participant)
Population: Safety Analysis set of subjects enrolled - Number of Patients with at least 1 event
Measure: Count of Participants; unit: Participants
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 13 | 12
Participants
  Number of Participants with Adverse Device Effects | 0 | 0
  Number of Participants with Serious Adverse Device Effects | 0 | 0

3. Other Pre Specified Outcome: Mean Change in IOP Through Week 24 Compared to Baseline
Description: Change from baseline in intraocular pressure as measured by applanation tonometry or standard IOP measuring devices
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: Efficacy Evaluable Population of participants with completed administration of trial treatment and at least one post baseline measurement in the study eye
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 10 | 10
mmHg
  Mean Change in IOP from Baseline at Week 4 | 1.6 (5.0) | 1.0 (2.5)
  Mean Change in IOP from Baseline at Week 12: number analyzed (Participants) | 8 | 6
  Mean Change in IOP from Baseline at Week 12 | 1.6 (2.9) | -0.2 (4.4)
  Mean Change in IOP from Baseline at Week 24: number analyzed (Participants) | 4 | 3
  Mean Change in IOP from Baseline at Week 24 | 1.3 (2.1) | 2.0 (3.6)

4. Other Pre Specified Outcome: Mean Change in Central Subfield Thickness (CST) at Study Visits Through Week 24 Compared to Baseline
Description: Change from Baseline in central subfield thickness (CST), to image the macular edema in the circular area 1 mm in diameter centered around the fovea. CST was measured using spectral domain optical coherence tomography (SD-OCT) and was read at the site. A negative change from baseline value represents a reduction in macular edema.
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 10 | 10
µm
  Mean Change in Central subfield thickness (CST) at Week 4 compared to baseline: number analyzed (Participants) | 8 | 9
  Mean Change in Central subfield thickness (CST) at Week 4 compared to baseline | -112.3 (136.2) | -172.0 (234.1)
  Mean Change in Central subfield thickness (CST) at Week 12 compared to baseline: number analyzed (Participants) | 7 | 4
  Mean Change in Central subfield thickness (CST) at Week 12 compared to baseline | -63.3 (71.4) | -132.8 (133.6)
  Mean Change in Central subfield thickness (CST) at Week 24 compared to baseline: number analyzed (Participants) | 4 | 3
  Mean Change in Central subfield thickness (CST) at Week 24 compared to baseline | -62.5 (45.0) | -127.7 (198.2)

5. Other Pre Specified Outcome: Mean Change in Best-Corrected Visual Acuity at Study Visits Through Week 24 Compared to Baseline
Description: Best corrected visual acuity (BCVA) using the ETDDRS methodology) with assessment starting at a distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
Time Frame: Baseline, Week 4, Week 12, and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 10 | 10
ETDRS letters
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at Week 4 Compared to Baseline: number analyzed (Participants) | 8 | 9
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at Week 4 Compared to Baseline | 4.5 (4.7) | 10.6 (10.0)
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at Week 12 Compared to Baseline: number analyzed (Participants) | 7 | 4
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at Week 12 Compared to Baseline | 0.9 (6.0) | 9.0 (9.6)
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at a Week 24 Compared to Baseline: number analyzed (Participants) | 4 | 3
  Mean Change in Best-Corrected Visual Acuity (ETDRS) at a Week 24 Compared to Baseline | 4.8 (11.8) | 11.0 (11.5)

6. Other Pre Specified Outcome: Number of Participants With Change in Best Corrected Visual Acuity (BCVA) Categorized as at Least 5, 10, and 15 Letter Gain Compared to Baseline at Study Visits Through Week 24
Description: Measure Description: Best corrected visual acuity (BCVA) at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
  The Outcome Measure provides the number of participants, who have at least a 5, 10, or 15 letter BCVA gain at the respective study visit compared to their baseline BCVA assessment
Time Frame: Baseline, Week 4, Week12, and Week 24
Population: Best corrected visual acuity (BCVA) at a starting distance of 4 meters. The BCVA letter score ranges from 0 to 100 (best score attainable), with a higher score indicating better visual acuity.
Measure: Count of Participants; unit: Participants
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
Number analyzed (Participants) | 10 | 10
Participants
  Week 4 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 8 | 9
  Week 4 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline | 5 | 6
  Week 12 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 7 | 4
  Week 12 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline | 1 | 3
  Week 24 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 4 | 3
  Week 24 At Least 5 Letter Gain in BCVA (ETDRS) compared to baseline | 2 | 2
  Week 4 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 8 | 9
  Week 4 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline | 1 | 5
  Week 12 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 7 | 4
  Week 12 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline | 1 | 2
  Week 24 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 4 | 3
  Week 24 At Least 10 Letter Gain in BCVA (ETDRS) compared to baseline | 2 | 2
  Week 4 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 8 | 9
  Week 4 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline | 0 | 3
  Week 12 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 7 | 4
  Week 12 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline | 0 | 1
  Week 24 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline: number analyzed (Participants) | 4 | 3
  Week 24 At Least 15 Letter Gain in BCVA (ETDRS) compared to baseline | 2 | 1

ADVERSE EVENTS:
Time Frame: Day 0 up to Week 24. The maximum interval of trial participation was 24 weeks, but per protocol participants ended their trial participation starting at Week 4, if they met criteria for follow-on therapy to treat Diabetic Macular Edema (DME)
Arm/Group | Suprachoroidal Triamcinolone Acetonide 2.4mg | Suprachoroidal Triamcinolone Acetonide 4.0mg
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 12/13 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Suprachoroidal Triamcinolone Acetonide 2.4mg (N=13) | Suprachoroidal Triamcinolone Acetonide 4.0mg (N=12)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blepharitis - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Cataract - Study Eye (Eye disorders) | 1 (1) | 1 (1)
Conjunctival Oedema - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage - Study Eye (Eye disorders) | 8 (8) | 7 (7)
Conjunctival hyperemia - Study Eye (Eye disorders) | 3 (3) | 1 (1)
Corneal abrasion - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Episcleritis - Study Eye (Eye disorders) | 1 (1) | 0 (0)
Eyelid Ptosis - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Eye Pain - Study Eye (Eye disorders) | 2 (2) | 4 (4)
Retinal Hemorrhage - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Vitreous Detachment - Study eye (Eye disorders) | 0 (0) | 1 (1)
Vitreous hemorrhage - Study Eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Treatment Failure (Trial procedure not completed in the study eye) (General disorders) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3)
Conjunctival laceration - Study Eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Underdose - Treatment Study Eye (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wrong route - Treatment Study Eye (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraocular pressure increased - Study Eye (Investigations) | 1 (1) | 0 (0)
Prostate-specific antigen increased (Investigations) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostate hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vitreous Detachment - Fellow Eye (Eye disorders) | 0 (0) | 1 (1)
Cataract - Fellow Eye (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/62/NCT05512962/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/62/NCT05512962/SAP_001.pdf